CLINICAL TRIAL: NCT03044808
Title: Randomized Double Blind Prospective Investigation of the Effect of Intravenous Lidocaine Infusion on Postoperative Pain Treatment and Bowel Function in Robotic Bowel Surgery
Brief Title: Investigation of the Effect of Intravenous Lidocaine Infusion on Postoperative Pain Treatment and Bowel Function in Robotic Bowel Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Jan Herzog, M.D., Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13.024; 2014-003466-25 (EudraCT Number)
Record Dates: First submitted 2017-02-03; First posted 2017-02-07 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Opioid Use
MeSH Terms: interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: 2 randomized groups, one getting lidocaine and the other getting saline
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Pharmacy provides the research medicine, it is not possible to see a difference. The envelopes are "encrypted". The randomization will only be broken in the end.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lidocain (Experimental): Patient gets the experimental treatment with IV lidocain 0,5mg/ml, 1,5mg/kg bolus before induction of anesthesia, after that infusion of 1,5mg/kg/h is started and continued until 2 hours after end of surgery.
  Interventions: Drug: Lidocaine
- Control (Placebo Comparator): Patients get the same amount in ml and duration as if it was the experimental arm. Only in this arm it is isotonic saline instead.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Lidocaine
  Arms: Lidocain
Drug: Saline
  Arms: Control

SUMMARY:
Single center double blind randomised controlled trial. 60 subjects. Giving lidocaine IV or saline to patients due to robot assisted colorectal surgery. Primary outcome is cumulative morphine consumption at 24 hours.

DETAILED DESCRIPTION:
Prospective double blind randomised controlled trial. The investigators are giving lidocaine IV or saline to 60 patients undergoing robot assisted colorectal surgery. Blinding and randomization is done by the hospital pharmacy. Both groups get otherwise the same treatment and a IV PCA (patient controlled administration) morphine pump for objectivisation of opioid consumption. Other outcome measures are NRS (numerical rating score) pain score, PONV (postoperative nausea and vomiting), use of antiemetics and opioid consumption up to 72 hours.

ELIGIBILITY:
Inclusion Criteria:

* all patients due to robotic laparoscopic colorectal surgery, > 18years of age, danish speaking

Exclusion Criteria:

* allergy to lidocain or amid local analgetics, atrioventricular blok, liver- and/or kidney failure, chronic use of opioids or NSAIDS, pregnancy, breastfeeding women, treatment with betablockers, porphyria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-02-02 (Actual); Primary Completion 2017-04-19 (Actual); Study Completion 2017-04-19 (Actual)

PRIMARY OUTCOMES:
Reduction in morphine consumption | over the first 24 hours
  PCA morphine added to PN (per necessitae) morphine, cumulated

SECONDARY OUTCOMES:
PONV | up to 72 hours
  Postoperative nausea and vomiting - patient is asked
Reduction in morphine consumption | over the first 72hours
  PCA morphine added to PN morphine, cumulated
Use of antiemetics postoperative | first 72 hours
Time to bowel function | first 72 hours
  time to flatus or defecation or function of bowel stoma
time to discharge | up to 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Odense Universitetshospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Herzog J, Schou M, Jensen KM, Lauridsen JT, Jensen AG. A randomised controlled trial of lidocaine infusion on post-operative opioid consumption in patients undergoing robotic colorectal surgery. Dan Med J. 2020 Jan;67(1):A06190342. PMID 31908254